CLINICAL TRIAL: NCT04305496
Title: A Phase III Double-blind Randomised Study Assessing the Efficacy and Safety of Capivasertib + Fulvestrant Versus Placebo + Fulvestrant as Treatment for Locally Advanced (Inoperable) or Metastatic Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative (HR+/HER2-) Breast Cancer Following Recurrence or Progression On or After Treatment With an Aromatase Inhibitor
Brief Title: Capivasertib+Fulvestrant vs Placebo+Fulvestrant as Treatment for Locally Advanced (Inoperable) or Metastatic HR+/HER2- Breast Cancer
Acronym: CAPItello-291
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3615C00001; 2023-505042-25-00 (Registry Identifier: CTIS (EU)); 2019-003629-78 (EudraCT Number)
Record Dates: First submitted 2020-02-20; First posted 2020-03-12 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced (Inoperable) or Metastatic Breast Cancer
Keywords: Locally advanced (inoperable) or Metastatic Breast Cancer
MeSH Terms: interventions — Fulvestrant; capivasertib

STUDY DESIGN:
Intervention Model Description: Double-blind Randomised Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capivasertib + fulvestrant (Experimental): Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 of Weeks 1 and 3 of cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
  Capivasertib: 400 mg (2 oral tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 1 to 4 in each week of a 28-day treatment cycle.
  Interventions: Drug: Fulvestrant; Drug: Capivasertib
- Placebo + fulvestrant (Placebo Comparator): Fulvestrant: 2 intramuscular injections of 500 mg given on Day 1 of Weeks 1 and 3 of cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
  Placebo: 400 mg (2 oral tablets) BD given on an intermittent weekly dosing schedule. Dosed on Days 1 to 4 in each week of a 28-day treatment cycle.
  Interventions: Drug: Fulvestrant; Drug: Placebo

INTERVENTIONS:
Drug: Fulvestrant — Patients will be administered 500 mg (2 injections) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter
Drug: Capivasertib — 400 mg BD (2 tablets of 200 mg taken twice a day = total daily dose 800 mg) given on an intermittent weekly dosing schedule. Patients will be dosed on Days 1 to 4 in each week of a 28-day treatment cycle
  Arms: Capivasertib + fulvestrant
Drug: Placebo — Placebo to match 400 mg BD (2 tablets of placebo to match 200 mg taken twice daily = placebo to match total daily dose of 800 mg) given on an intermittent weekly dosing schedule. Patients will be dosed on Days 1 to 4 in each week of a 28-day treatment cycle
  Arms: Placebo + fulvestrant

SUMMARY:
Phase III, double-blind, randomised study assessing the efficacy of capivasertib + fulvestrant vs placebo + fulvestrant for the treatment of patients with locally advanced (inoperable) or metastatic HR+/HER2- breast cancer following recurrence or progression on or after AI therapy.

DETAILED DESCRIPTION:
Phase III, double-blind, randomised study assessing the efficacy of capivasertib + fulvestrant vs placebo + fulvestrant for the treatment of patients with locally advanced (inoperable) or metastatic Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative (HR+/HER2-) breast cancer following recurrence or progression on or after aromatase inhibitor (AI) therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females, pre- and/or post-menopausal, and adult males. Pre-menopausal (and peri-menopausal) women can be enrolled if amenable to treatment with an LHRH agonist. Patients are to have commenced concomitant treatment with LHRH agonist prior to or on Cycle 1, Day 1 and must be willing to continue on it for the duration of the study
2. Histologically confirmed HR+/HER2- breast cancer determined from the most recent tumour sample (primary or metastatic), as per the American Society of Clinical Oncology and College of American Pathologists guideline recommendations. To fulfil the requirement of HR+ disease, a breast cancer must express ER with or without co-expression of progesterone receptor.
3. Metastatic or locally advanced disease with radiological or objective evidence of recurrence or progression (the cancer should have shown progression during or after most recent therapy); locally advanced disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible)
4. ECOG/WHO PS: 0-1
5. Patients are to have received treatment with an AI (aromatase inhibitor) containing regimen (single agent or in combination) and have:

   1. Radiological evidence of breast cancer recurrence or progression while on, or within 12 months of the end of (neo)adjuvant treatment with an AI, OR
   2. Radiological evidence of progression while on prior AI administered as a treatment line for locally advanced or metastatic breast cancer (this does not need to be the most recent therapy)
6. Patients must have measurable disease according to RECIST 1.1 and/or at least 1 lytic or mixed (lytic + sclerotic) bone lesion that can be assessed by CT or MRI; patients with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible
7. FFPE tumour sample from primary/recurrent cancer for central testing

Exclusion Criteria:

1. Symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine therapy per the investigator's best judgement
2. More than 2 lines of endocrine therapy for inoperable locally advanced or metastatic disease
3. More than 1 line of chemotherapy for inoperable locally advanced or metastatic disease. Adjuvant and neoadjuvant chemotherapy are not classed as lines of chemotherapy for advanced breast cancer
4. Prior treatment with any of the following:

   1. AKT, PI3K and mTOR inhibitors
   2. Fulvestrant, and other SERDs
   3. Any other chemotherapy, immunotherapy, immunosuppressant medication (other than corticosteroids) or anticancer agents within 3 weeks prior to study treatment initiation.
   4. Potent inhibitors or inducers of CYP3A4 within 2 weeks prior to the first dose of study treatment (3 weeks for St John's wort) or drugs that are sensitive to CYP3A4 inhibition within 1 week prior to study treatment initiation.
5. Radiotherapy with a wide field of radiation up to 4 weeks before study treatment initiation (capivasertib/placebo) and/or radiotherapy with a limited field of radiation for palliation up to 2 weeks before study treatment initiation (capivasertib/placebo)
6. With the exception of alopecia, any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment
7. Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring steroids up to 4 weeks before study treatment initiation
8. Any of the following cardiac criteria:

   1. Mean resting QT interval corrected by Fridericia's formula (QTcF) >470 msec obtained from 3 consecutive ECGs
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (eg, complete left bundle branch block, third degree heart block)
   3. Any factors that increase the risk of corrected QT interval (QTc) prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval
   4. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association (NYHA) grade ≥2
   5. Uncontrolled hypotension - systolic blood pressure <90 mmHg and/or diastolic blood pressure <50 mmHg
   6. Cardiac ejection fraction outside institutional range of normal or <50% (whichever is higher) as measured by echocardiogram (or multiple-gated acquisition [MUGA] scan if an echocardiogram cannot be performed or is inconclusive)
9. Clinically significant abnormalities of glucose metabolism as defined by any of the following:

   1. Patients with diabetes mellitus type 1 or diabetes mellitus type 2 requiring insulin treatment
   2. HbA1c ≥8.0% (63.9 mmol/mol)
10. Known abnormalities in coagulation such as bleeding diathesis, or treatment with anticoagulants precluding intramuscular injections of fulvestrant or LHRH agonist (if applicable)
11. Currently pregnant (confirmed with positive pregnancy test) or breast-feeding

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2026-06-22 (Estimated)

CONTACTS AND LOCATIONS:
Locations (179):
- United States (22):
  - Research Site, Gilbert, Arizona
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Whittier, California
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Westwood, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Paramus, New Jersey
  - Research Site, Farmington, New Mexico
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Midlothian, Virginia
  - Research Site, Puyallup, Washington
- Argentina (5):
  - Research Site, Berazategui
  - Research Site, Buenos Aires
  - Research Site, La Rioja
  - Research Site, Rosario
  - Research Site, Viedma
- Australia (12):
  - Research Site, Adelaide
  - Research Site, Ballarat
  - Research Site, Birtinya
  - Research Site, Box Hill
  - Research Site, Concord
  - Research Site, Kurralta Park
  - Research Site, North Sydney
  - Research Site, Orange
  - Research Site, Ringwood East
  - Research Site, South Brisbane
  - Research Site, Waratah
  - Research Site, Wendouree
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Namur
  - Research Site, Wilrijk
- Canada (4):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Kingston, Ontario
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
- China (21):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chongqing
  - Research Site, Dalian
  - Research Site, Foshan
  - Research Site, Gongshu District
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nantong
  - Research Site, Neijiang
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- France (9):
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Metz
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Pringy
  - Research Site, Rouen
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (15):
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Gelsenkirchen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Mannheim
  - Research Site, Minden
  - Research Site, München
  - Research Site, Münster
  - Research Site, Paderborn
  - Research Site, Potsdam
- Hungary (5):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kecskemét
  - Research Site, Szekszárd
  - Research Site, Szolnok
- Israel (7):
  - Research Site, Afula
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
- Italy (11):
  - Research Site, Bergamo
  - Research Site, Candiolo
  - Research Site, Catanzaro
  - Research Site, Livorno
  - Research Site, Macerata
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Prato
  - Research Site, Roma
- Japan (18):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Kagoshima
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Ota-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Tsu
  - Research Site, Yokohama
- Peru (2):
  - Research Site, Arequipa
  - Research Site, Lima
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Olsztyn
  - Research Site, Warsaw
- Russia (4):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Sochi
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (15):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Hosp de Llobregat(Barcelona)
  - Research Site, Jaén
  - Research Site, La Laguna (Tenerife)
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Reus
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (8):
  - Research Site, Aberdeen
  - Research Site, Bournemouth
  - Research Site, Bristol
  - Research Site, Cardiff
  - Research Site, Cheltenham
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Turner NC, Oliveira M, Howell SJ, Dalenc F, Cortes J, Gomez Moreno HL, Hu X, Jhaveri K, Krivorotko P, Loibl S, Morales Murillo S, Okera M, Park YH, Sohn J, Toi M, Tokunaga E, Yousef S, Zhukova L, de Bruin EC, Grinsted L, Schiavon G, Foxley A, Rugo HS; CAPItello-291 Study Group. Capivasertib in Hormone Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2023 Jun 1;388(22):2058-2070. doi: 10.1056/NEJMoa2214131. PMID 37256976
- [Derived] Turner NC, Oliveira M, Howell SJ, Dalenc F, Cortes J, Gomez HL, Hu X, Jhaveri K, Krivorotko P, Loibl S, Murillo SM, Park YH, Sohn JH, Toi M, Tokunaga E, Yousef S, Zhukova L, de Bruin E, Grinsted L, Schiavon G, Foxley A, Rugo HS. A plain language summary of the CAPItello-291 study: Capivasertib in hormone receptor-positive advanced breast cancer. Future Oncol. 2024;20(37):2901-2913. doi: 10.1080/14796694.2024.2390791. Epub 2024 Sep 16. PMID 39283299
- [Derived] Oliveira M, Rugo HS, Howell SJ, Dalenc F, Cortes J, Gomez HL, Hu X, Toi M, Jhaveri K, Krivorotko P, Loibl S, Morales Murillo S, Okera M, Nowecki Z, Park YH, Sohn JH, Tokunaga E, Yousef S, Zhukova L, Fulford M, Andrews H, Wadsworth I, D'Cruz C, Turner NC; CAPItello-291 study group. Capivasertib and fulvestrant for patients with hormone receptor-positive, HER2-negative advanced breast cancer (CAPItello-291): patient-reported outcomes from a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2024 Sep;25(9):1231-1244. doi: 10.1016/S1470-2045(24)00373-5. PMID 39214106
- [Derived] Dilawari A, Buturla J, Osgood C, Gao X, Chen W, Ricks TK, Schaefer T, Avasarala S, Reyes Turcu F, Pathak A, Kalavar S, Bhatnagar V, Collazo J, Rahman NA, Mixter B, Tang S, Pazdur R, Kluetz P, Amiri-Kordestani L. US Food and Drug Administration Approval Summary: Capivasertib With Fulvestrant for Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Locally Advanced or Metastatic Breast Cancer With PIK3CA/AKT1/PTEN Alterations. J Clin Oncol. 2024 Dec;42(34):4103-4113. doi: 10.1200/JCO.24.00427. Epub 2024 Aug 19. PMID 39159418
- See also: CSP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3615C00001&attachmentIdentifier=ea4213cd-5dc8-499b-9f8d-12cad4e051f5&fileName=csp-redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3615C00001&attachmentIdentifier=0bdafe79-ad18-464d-8706-02a02a1282cf&fileName=sap-redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3615C00001&attachmentIdentifier=0b3062da-fd98-4449-a963-453cef8e7e25&fileName=csr_synopsis-redacted.pdf&versionIdentifier=
- See also: CSR Synopsis China Cohort — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3615C00001&attachmentIdentifier=f974c655-0157-499e-bdb3-b362272db8a5&fileName=CSR_Synopsis_China_Cohort.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 708 participants in Global cohort (out of 818 participants in Global and China cohorts) were randomized to treatment. An additional 110 participants were enrolled into the China cohort only.
Pre-assignment Details: A total of 818 participants were enrolled in the study. However, 24 participants were in both the Global and China cohorts.
Groups:
- Capivasertib + Fulvestrant: Capivasertib: 400 mg twice daily (2 tablets of 200 mg taken orally twice daily; total daily dose 800 mg) given on an intermittent weekly dosing schedule (4 days on/3 days off).
  Fulvestrant: 500 mg (2 intramuscular injections of 250 mg/5 mL solution) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
- Placebo + Fulvestrant: Placebo: Placebo tablets matching capivasertib. 400 mg twice daily (2 tablets of 200 mg taken orally twice daily; total daily dose 800 mg) given on an intermittent weekly dosing schedule (4 days on/3 days off).
  Fulvestrant: 500 mg (2 intramuscular injections of 250 mg/5 mL solution) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
Period: Global Cohort
Arm/Group | Capivasertib + Fulvestrant | Placebo + Fulvestrant
Started | 355 | 353
Completed | 63 (Participants ongoing capivasertib/placebo at data cut-off) | 43 (Participants ongoing capivasertib/placebo at data cut-off)
Not Completed | 292 | 310
Not completed — Withdrawal by Subject | 13 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Subjective disease progression | 16 | 17
Not completed — Condition under investigation worsened | 209 | 273
Not completed — Protocol Violation | 2 | 0
Not completed — Adverse Event | 44 | 6
Not completed — Death | 3 | 2
Not completed — Any reason not specifically recorded | 4 | 5
Period: China Cohort
Arm/Group | Capivasertib + Fulvestrant | Placebo + Fulvestrant
Started | 71 (An additional 110 participants were enrolled into the China cohort only; 24 participants were in both the Global and China cohorts.) | 63 (An additional 110 participants were enrolled into the China cohort only; 24 participants were in both the Global and China cohorts.)
Completed | 18 (Participants ongoing capivasertib/placebo at data cut-off) | 10 (Participants ongoing capivasertib/placebo at data cut-off)
Not Completed | 53 | 53
Not completed — Any reason not specifically recorded | 1 | 1
Not completed — Adverse Event | 8 | 2
Not completed — Condition under investigation worsened | 40 | 47
Not completed — Subjective disease progression | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set. 24 participants (16 participants in the capivasertib arm and 8 participants in the placebo arm) were included in both the Global and China cohorts.
Groups:
- Capivasertib + Fulvestrant (Global + China Cohort): Capivasertib: 400 mg twice daily (2 tablets of 200 mg taken orally twice daily; total daily dose 800 mg) given on an intermittent weekly dosing schedule (4 days on/3 days off).
  Fulvestrant: 500 mg (2 intramuscular injections of 250 mg/5 mL solution) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
- Placebo + Fulvestrant (Global Cohort + China Cohort ): Placebo: Placebo tablets matching capivasertib. 400 mg twice daily (2 tablets of 200 mg taken orally twice daily; total daily dose 800 mg) given on an intermittent weekly dosing schedule (4 days on/3 days off).
  Fulvestrant: 500 mg (2 intramuscular injections of 250 mg/5 mL solution) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
- Total: Total of all reporting groups
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global Cohort + China Cohort ) | Total
Number analyzed (Participants) | 410 | 408 | 818
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The results are presented by Global cohort and by China cohort
  years
    Global cohort: number analyzed (Participants) | 355 | 353 | 708
    Global cohort | 58.6 (11.25) | 57.4 (11.91) | 58.0 (11.59)
    China cohort: number analyzed (Participants) | 71 | 63 | 134
    China cohort | 54.7 (10.66) | 55.0 (10.60) | 54.8 (10.59)
Age, Customized [Count of Participants; unit: Participants] — Age at Screening Population: Overall population
  Participants
    Global cohort: number analyzed (Participants) | 355 | 353 | 708
    Global cohort: <50 years | 76 | 99 | 175
    Global cohort: >=50-<65 years | 164 | 152 | 316
    Global cohort: >=65-<75 years | 91 | 76 | 167
    Global cohort: >=75 years | 24 | 26 | 50
    China cohort: number analyzed (Participants) | 71 | 63 | 134
    China cohort: <50 years | 19 | 24 | 43
    China cohort: >=50-<65 years | 39 | 21 | 60
    China cohort: >=65-<75 years | 12 | 18 | 30
    China cohort: >=75 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort
  Participants
    Global cohort: number analyzed (Participants) | 355 | 353 | 708
    Global cohort: Female | 352 | 349 | 701
    Global cohort: Male | 3 | 4 | 7
    China cohort: number analyzed (Participants) | 71 | 63 | 134
    China cohort: Female | 71 | 62 | 133
    China cohort: Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort
  Participants
    Global cohort: number analyzed (Participants) | 355 | 353 | 708
    Global cohort: Hispanic or Latino | 31 | 31 | 62
    Global cohort: Not Hispanic or Latino | 323 | 322 | 645
    Global cohort: Unknown or Not Reported | 1 | 0 | 1
    China cohort: number analyzed (Participants) | 71 | 63 | 134
    China cohort: Hispanic or Latino | 0 | 0 | 0
    China cohort: Not Hispanic or Latino | 69 | 61 | 130
    China cohort: Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The results are presented by Global cohort and by China cohort
  Participants
    Global cohort: number analyzed (Participants) | 355 | 353 | 708
    Global cohort: American Indian or Alaska Native | 2 | 2 | 4
    Global cohort: Asian | 95 | 94 | 189
    Global cohort: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Global cohort: Black or African American | 4 | 4 | 8
    Global cohort: White | 201 | 206 | 407
    Global cohort: More than one race | 0 | 0 | 0
    Global cohort: Unknown or Not Reported | 52 | 47 | 99
    China cohort: number analyzed (Participants) | 71 | 63 | 134
    China cohort: American Indian or Alaska Native | 0 | 0 | 0
    China cohort: Asian | 69 | 61 | 130
    China cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    China cohort: Black or African American | 0 | 0 | 0
    China cohort: White | 0 | 0 | 0
    China cohort: More than one race | 0 | 0 | 0
    China cohort: Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival: Overall Population (Months) in the Global Cohort
Description: Progression free survival (PFS), defined as the time from randomization until progression per RECIST v1.1, as assessed by the investigator at the local site, or death due to any cause, in the global cohort.
  Participants who discontinue treatment prior to progression should continue to be scanned until progression.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of the longest diameter of target lesions (short axis diameter used for lymph nodes), or clinically significant increase in a non-target lesion, or the appearance of a new lesion(s).
Time Frame: Assessed every 8 weeks for the first 18 months and every 12 weeks thereafter, from randomization to radiological progression.
Population: Overall population in the global cohort
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo + Fulvestrant (Global + China Cohort): Placebo: Placebo tablets matching capivasertib. 400 mg twice daily (2 tablets of 200 mg taken orally twice daily; total daily dose 800 mg) given on an intermittent weekly dosing schedule (4 days on/3 days off).
  Fulvestrant: 500 mg (2 intramuscular injections of 250 mg/5 mL solution) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global + China Cohort)
Number analyzed (Participants) | 355 | 353
Months | 7.2 [5.5 to 7.4] | 3.6 [2.8 to 3.7]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort) vs Placebo + Fulvestrant (Global + China Cohort); Test type: Superiority; p < 0.001, Stratified log rank test; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.51 to 0.71]

2. Primary Outcome: Progression Free Survival: Overall Population (Percentage) in the Global Cohort
Description: Progression free survival (PFS), defined as the time from randomization until progression per RECIST v1.1, as assessed by the investigator at the local site, or death due to any cause.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of the longest diameter of target lesions (short axis diameter used for lymph nodes), or clinically significant increase in a non-target lesion, or the appearance of a new lesion(s).
  Participants who discontinue treatment prior to progression should continue to be scanned until progression.
  Kaplan-Meier estimate was used.
Time Frame: as for outcome 1
Population: Overall population in the Global Cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global + China Cohort)
Number analyzed (Participants) | 355 | 353
Percentage of participants
  PFS rate at 6 months | 51.8 [46.4 to 57.0] | 32.0 [27.0 to 37.0]
  PFS rate at 9 months | 40.9 [35.6 to 46.1] | 24.4 [19.9 to 29.1]
  PFS rate at 12 months | 28.5 [23.7 to 33.5] | 18.4 [14.4 to 22.8]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort); Test type: Superiority; p < 0.001, Stratified log rank test; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.51 to 0.71]

3. Primary Outcome: Progression Free Survival: Altered Population (Months) in the Global Cohort
Description: Progression free survival (PFS), defined as the time from randomization until progression per RECIST v1.1, as assessed by the investigator at the local site, or death due to any cause.
Time Frame: Assessed every 8 weeks for the first 2 years following objective disease progression or treatment discontinuation and then every 12 weeks.
Population: Altered population in the Global Cohort
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global + China Cohort)
Number analyzed (Participants) | 155 | 134
Months | 7.3 [5.5 to 9.0] | 3.1 [2.0 to 3.7]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort) vs Placebo + Fulvestrant (Global + China Cohort); Test type: Superiority; p < 0.001, Stratified log-rank test; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.38 to 0.65]

4. Primary Outcome: Progression Free Survival: Altered Population (Percentage) in the Global Cohort
Description: Progression free survival (PFS), defined as the time from randomization until progression per RECIST v1.1, as assessed by the investigator at the local site, or death due to any cause.
  Kaplan-Meier estimate was used.
Time Frame: as for outcome 3
Population: Altered population in the Global Cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global + China Cohort)
Number analyzed (Participants) | 155 | 134
Percentage of participants
  PFS rate at 6 months | 53.4 [45.1 to 60.9] | 29.6 [21.9 to 37.7]
  PFS rate at 9 months | 42.0 [34.0 to 49.7] | 21.6 [14.9 to 29.1]
  PFS rate at 12 months | 28.2 [21.2 to 35.6] | 15.8 [10.0 to 22.7]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort) vs Placebo + Fulvestrant (Global + China Cohort); Test type: Superiority; p < 0.001, Stratified log-rank test; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.38 to 0.65]

5. Primary Outcome: Progression Free Survival: Overall Population (Months) in the China Cohort
Description: Progression free survival (PFS), defined as the time from randomization until progression per RECIST v1.1, as assessed by the investigator at the local site, or death due to any cause, in the global cohort.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of the longest diameter of target lesions (short axis diameter used for lymph nodes), or clinically significant increase in a non-target lesion, or the appearance of a new lesion(s).
  Participants who discontinue treatment prior to progression should continue to be scanned until progression.
Time Frame: as for outcome 1
Population: Full analysis set in the China cohort
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Placebo + Fulvestrant (China Cohort): Placebo: Placebo tablets matching capivasertib. 400 mg twice daily (2 tablets of 200 mg taken orally twice daily; total daily dose 800 mg) given on an intermittent weekly dosing schedule.Fulvestrant: 500 mg (2 intramuscular injections of 250 mg/5 mL solution) on Day 1 of Weeks 1 and 3 of Cycle 1, and then on Day 1, Week 1 of each cycle thereafter.
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (China Cohort)
Number analyzed (Participants) | 71 | 63
Months | 6.9 [5.4 to 9.2] | 2.8 [1.9 to 3.9]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort); Test type: Superiority; p < 0.001, Stratified log rank test; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.34 to 0.76]

6. Primary Outcome: Progression Free Survival: Overall Population (Percentage) in the China Cohort
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Full analysis set in the China cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (China Cohort)
Number analyzed (Participants) | 71 | 63
Percentage of participants
  PFS rate at 6 months | 53.9 [41.3 to 65.0] | 24.5 [14.6 to 35.8]
  PFS rate at 9 months | 40.9 [28.8 to 52.5] | 24.5 [14.6 to 35.8]
  PFS rate at 12 months | 29.6 [18.6 to 41.4] | 19.1 [10.3 to 29.9]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort); Test type: Superiority; p < 0.001, Stratified log rank test; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.34 to 0.76]

7. Primary Outcome: Progression Free Survival: Altered Population (Months) in the China Cohort
Description: as for outcome 3
Time Frame: as for outcome 3
Population: Altered subgroup full analysis set in the China cohort
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global + China Cohort)
Number analyzed (Participants) | 71 | 63
Months | 5.7 [3.8 to 8.0] | 1.9 [1.8 to 3.7]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort); Test type: Superiority; p = 0.016, Stratified log rank test; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.19 to 0.85]

8. Primary Outcome: Progression Free Survival: Altered Population (Percentage) in the China Cohort
Description: Progression free survival (PFS), defined as the time from randomization until progression per RECIST v1.1, as assessed by the investigator at the local site, or death due to any cause
  Kaplan-Meier estimate was used.
Time Frame: as for outcome 3
Population: Altered subgroup full analysis set in the China cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capivasertib + Fulvestrant (Global + China Cohort) | Placebo + Fulvestrant (Global + China Cohort)
Number analyzed (Participants) | 71 | 63
Percentage of participants
  PFS rate at 6 months | 46.3 [25.1 to 65.1] | 14.3 [3.6 to 32.1]
  PFS rate at 9 months | 23.1 [8.5 to 42.0] | 14.3 [3.6 to 32.1]
  PFS rate at 12 months | 6.9 [0.6 to 24.9] | 14.3 [3.6 to 32.1]
Statistical Analysis 1: Comparison: Capivasertib + Fulvestrant (Global + China Cohort); Test type: Superiority; p = 0.016, Stratified log rank test; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.19 to 0.85]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from time of signature of the informed consent form, throughout the treatment period and including the 30-day follow-up period after discontinuation of study drug. Only treatment emergent AEs are presented.
Description: Full analysis set is included for mortality rate, but safety analysis set is included other SAEs/nonserious AEs.
  An AE was development of any untoward medical occurrence/deterioration of preexisting medical occurrence in a participant administered medicinal product, which did not necessarily have a causal relationship with treatment, including SAEs and non-serious AEs. AEs of special interest were identified and actively monitored.
  Only fatal AEs are presented for all-cause mortality.
Groups:
- Capi (Global Cohort); Placebo (Global Cohort); Capi (China Cohort); Placebo (China Cohort): Description (Arm-group)
Arm/Group | Capi (Global Cohort) | Placebo (Global Cohort) | Capi (China Cohort) | Placebo (China Cohort)
All-Cause Mortality (participants affected / at risk) | 4/355 | 1/350 | 1/71 | 0/62
Serious Adverse Events (participants affected / at risk) | 57/355 | 28/350 | 20/71 | 3/62
Other Adverse Events (participants affected / at risk) | 334/355 | 255/350 | 67/71 | 52/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capi (Global Cohort) (N=355) | Placebo (Global Cohort) (N=350) | Capi (China Cohort) (N=71) | Placebo (China Cohort) (N=62)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 3 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2 | 2 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Device intolerance (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Visceral pain (General disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Bacterial colitis (Infections and infestations) | 1 | 0 | 0 | 0
Bone tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis b reactivation (Infections and infestations) | 1 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0 | 0
Injection site abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 2 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 3 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capi (Global Cohort) (N=355) | Placebo (Global Cohort) (N=350) | Capi (China Cohort) (N=71) | Placebo (China Cohort) (N=62)
Dysgeusia (Nervous system disorders) | 21 | 4 | 1 | 1
Headache (Nervous system disorders) | 60 | 43 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 21 | 9 | 4 | 0
Insomnia (Psychiatric disorders) | 22 | 21 | 5 | 1
Proteinuria (Renal and urinary disorders) | 7 | 5 | 12 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 2 | 6
Constipation (Gastrointestinal disorders) | 28 | 29 | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 23 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 15 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 255 | 70 | 43 | 7
Erythema (Skin and subcutaneous tissue disorders) | 6 | 2 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 44 | 23 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 77 | 15 | 21 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 52 | 9 | 18 | 2
Hot flush (Vascular disorders) | 18 | 19 | 0 | 0
Hypertension (Vascular disorders) | 18 | 13 | 5 | 1
Dry mouth (Gastrointestinal disorders) | 19 | 9 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 18 | 7 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 7 | 1 | 6 | 2
Nausea (Gastrointestinal disorders) | 122 | 53 | 10 | 2
Anaemia (Blood and lymphatic system disorders) | 37 | 16 | 22 | 11
Stomatitis (Gastrointestinal disorders) | 51 | 17 | 9 | 0
Vomiting (Gastrointestinal disorders) | 70 | 15 | 7 | 3
Asthenia (General disorders) | 45 | 36 | 3 | 1
Fatigue (General disorders) | 73 | 45 | 3 | 2
Malaise (General disorders) | 10 | 7 | 3 | 8
Pyrexia (General disorders) | 32 | 13 | 16 | 3
Covid-19 (Infections and infestations) | 21 | 10 | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 4 | 1
Urinary tract infection (Infections and infestations) | 35 | 23 | 15 | 12
Alanine aminotransferase increased (Investigations) | 32 | 30 | 13 | 21
Aspartate aminotransferase increased (Investigations) | 33 | 33 | 10 | 18
Blood alkaline phosphatase increased (Investigations) | 13 | 12 | 6 | 7
Blood bilirubin increased (Investigations) | 2 | 4 | 4 | 1
Blood cholesterol increased (Investigations) | 1 | 5 | 6 | 4
Blood creatinine increased (Investigations) | 16 | 2 | 7 | 2
Blood thyroid stimulating hormone increased (Investigations) | 5 | 4 | 8 | 5
Blood urea increased (Investigations) | 2 | 2 | 4 | 0
Electrocardiogram qt prolonged (Investigations) | 3 | 0 | 5 | 0
Gamma-glutamyltransferase increased (Investigations) | 12 | 3 | 5 | 4
Glucose urine present (Investigations) | 1 | 0 | 4 | 0
Glycosylated haemoglobin increased (Investigations) | 5 | 0 | 13 | 3
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 5 | 1
Lymphocyte count decreased (Investigations) | 6 | 3 | 6 | 3
Neutrophil count decreased (Investigations) | 9 | 8 | 14 | 4
Weight decreased (Investigations) | 12 | 8 | 17 | 3
White blood cell count decreased (Investigations) | 6 | 4 | 15 | 5
White blood cells urine positive (Investigations) | 0 | 0 | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 59 | 22 | 8 | 3
Sinus tachycardia (Cardiac disorders) | 4 | 1 | 5 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 | 3 | 8 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 56 | 13 | 41 | 11
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 3 | 16 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 6 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 3 | 8 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 1 | 8 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 2 | 18 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 2 | 6 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 38 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 24 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 18 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 22 | 4 | 2

LIMITATIONS AND CAVEATS:
There were 24 participants who were included in both the global cohort and China cohort which gives a total of 818 participants instead of a total of 842 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT04305496/Prot_003.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT04305496/SAP_001.pdf